CLINICAL TRIAL: NCT00422916
Title: Evaluation of the Intervention Program "Obeldicks Light" for Overweight Children and Adolescents
Brief Title: Treatment of Overweight Children and Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Witten/Herdecke (Other)
Collaborators: University of Bremen (Other)
Responsible Party: Principal Investigator, Thomas Reinehr, Head of Department of Pediatric Endocrinology, Diabetes, and Nutrition Medicine, University of Witten/Herdecke
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: GFEL011174505
Record Dates: First submitted 2007-01-16; First posted 2007-01-17 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Overweight
MeSH Terms: conditions — Overweight | interventions — Behavior Therapy

ARMS (2):
- intervention arm (Experimental): Lifestyle Intervention based on Nutrition Treatment, exercise Treatment and behavorial treatment
  Interventions: Behavioral: behavioral intervention
- waiting list (No Intervention): waiting 6 months for Intervention without any intervention

INTERVENTIONS:
Behavioral: behavioral intervention
  Arms: intervention arm

SUMMARY:
The intervention program "Obeldicks light" is developed for overweight children aged 8-16 years. This intervention is gender - and age specific.

The 6-month intervention is based on nutrition course, behaviour therapy and exercise therapy. The evaluation compromised quality of structure, process and results of the intervention. 300 participants in a randomised controlled group design will be evaluated at 4 time points: baseline, end of intervention, 6 months after end of intervention and 12 months after end of intervention.Primary outcome measure is change of weight status as standard deviation score of BMI. Drop-outs will be interviewed to improve the intervention.

ELIGIBILITY:
Inclusion Criteria:

* overweight children

Exclusion Criteria:

* primary disease

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2007-01; Primary Completion 2009-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
change of weight status | 6 months

SECONDARY OUTCOMES:
Change of eating and exercise behaviour | 6 months
change of quality of life | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Petra Kolip, Prof, Study Chair — University of Bremen, Germany
Locations (1):
- Vestische Youth Hospital, Datteln, Germany

REFERENCES:
- [Derived] Reinehr T, Bucksch J, Muller A, Finne E, Kolip P. 7-Year follow-up of a lifestyle intervention in overweight children: Comparison to an untreated control group. Clin Nutr. 2018 Oct;37(5):1558-1562. doi: 10.1016/j.clnu.2017.08.017. Epub 2017 Aug 24. PMID 28882396
- [Derived] Finne E, Reinehr T, Schaefer A, Winkel K, Kolip P. Health-related quality of life in overweight German children and adolescents: do treatment-seeking youth have lower quality of life levels? Comparison of a clinical sample with the general population using a multilevel model approach. BMC Public Health. 2013 Jun 8;13:561. doi: 10.1186/1471-2458-13-561. PMID 23759033
- [Derived] Finne E, Reinehr T, Schaefer A, Winkel K, Kolip P. Changes in self-reported and parent-reported health-related quality of life in overweight children and adolescents participating in an outpatient training: findings from a 12-month follow-up study. Health Qual Life Outcomes. 2013 Jan 2;11:1. doi: 10.1186/1477-7525-11-1. PMID 23281620
- [Derived] Reinehr T, Schaefer A, Winkel K, Finne E, Toschke AM, Kolip P. An effective lifestyle intervention in overweight children: findings from a randomized controlled trial on "Obeldicks light". Clin Nutr. 2010 Jun;29(3):331-6. doi: 10.1016/j.clnu.2009.12.010. Epub 2010 Jan 27. PMID 20106567